CLINICAL TRIAL: NCT01987193
Title: Feasibility Study of Tumor Blood Flow Measurement by Detection of Positron Activation Post Proton Therapy
Brief Title: Feasibility Study of Tumor Blood Flow Measurement by Detection of Positron Activation Post Proton Therapy (DS01)
Status: Terminated | Type: Observational
Why Stopped: Slow accrual; funding stopped
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: UFPTI 1214 - DS01
Record Dates: First submitted 2013-10-24; First posted 2013-11-19 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Brain Cancer; Prostate Cancer; Lung Cancer
Keywords: Proton radiation; tumor blood flow
MeSH Terms: conditions — Brain Neoplasms; Prostatic Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is the development of noninvasive (having no direct contact) detector and electronic system that will directly measure tumor blood flow rate.

ELIGIBILITY:
Inclusion Criteria:

Solid tumors in the intracranial, thoracic, or pelvic regions.

Exclusion Criteria: N/A

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at radiation oncology clinic
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Patients with hypoxic tumor identified by tumor blood flow measurement. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Su, PhD, Principal Investigator — University of Florida Proton Therapy Institute
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided